CLINICAL TRIAL: NCT00581542
Title: A Single Blinded Clinical Trial Comparing Polytrim Ophthalmic Solution and Moxifloxacin Ophthalmic Solution for Treatment of Conjunctivitis.
Brief Title: Moxifloxacin vs. Polytrim for Conjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Frank Gigliotti, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RSRB #17454
Record Dates: First submitted 2007-12-18; First posted 2007-12-27 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-12

CONDITIONS: Conjunctivitis
MeSH Terms: conditions — Conjunctivitis | interventions — Moxifloxacin; Polytrim eyedrops

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin Opthalmic solution (Active Comparator)
  Interventions: Drug: polytrim
- Polymyxin B-trimethoprim opthalmic solution (Active Comparator)
  Interventions: Drug: moxifloxacin

INTERVENTIONS:
Drug: moxifloxacin — 1-2 drops three times a day for 8-10 days.
  Arms: Polymyxin B-trimethoprim opthalmic solution
Drug: polytrim — 1-2 drops four times a day for 8-10 days.
  Arms: Moxifloxacin Opthalmic solution

SUMMARY:
The purpose of the study is to compare the effect of Polytrim Ophthalmic Solution and Moxifloxacin Ophthalmic Solution in treating your child's pink eye. Both these medications are approved by the Food and Drug Administration, for treatment of conjunctivitis. This study will investigate if both of the medications are equally good.

ELIGIBILITY:
Inclusion Criteria:

* 1 - 18 years of age with presumed bacterial conjunctivitis.

Exclusion Criteria:

* Previous antibiotics or to receive systemic antibiotic.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Gigliotti, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Polytrim Group: Randomization to polytrim : 1-2 drops four times a day for 8-10 days.
- Moxifloxin Group: Randomization to topical moxifloxacin 1-2 drops 3x/day for 8-10 days
Period: Overall Study
Arm/Group | Polytrim Group | Moxifloxin Group
Started | 62 | 62
Completed | 51 | 39
Not Completed | 11 | 23
Not completed — they met an exclusion criteria | 2 | 2
Not completed — Lost to Follow-up | 9 | 21

BASELINE CHARACTERISTICS:
Groups:
- Polytrim Ophthalmic Solution: randomization to topical polytrim
- Moxifloxacin Ophthalmic Solution: randomization to topical moxifloxacin
- Total: Total of all reporting groups
Arm/Group | Polytrim Ophthalmic Solution | Moxifloxacin Ophthalmic Solution | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: months] | 73.4 (50) | 70.3 (48) | 71.3 (49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 28 | 67
  Male | 23 | 34 | 57
Region of Enrollment [Number; unit: participants]
  United States | 62 | 62 | 124

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Normal Physical Examination of the Eye
Time Frame: 10 days
Measure: Number; unit: participants
Arm/Group | Polytrim Arm | Moxifloxacin
Number analyzed (Participants) | 51 | 39
participants | 49 | 37

2. Secondary Outcome: Number of Participants With a Negative Bacterial Culture
Description: Conjunctival swab specimens were inoculated onto tryptic soy agar with 5% sheep blood and GC II agar supplemented with hemoglobin and isovialex with incubation at 35 degrees C in ambient air supplemented with 5% carbon dioxide for 48 hours. S pneumoniae, H influenzai and M Catarrhalis were identified.
Time Frame: 10 days
Population: Only participants who were culture positive at baseline were tested at day 10. 20 participants were negative at baseline in the polytrim group and 11 participants were negative in the moxifloxin group.
Measure: Number; unit: participants
Arm/Group | Moxifloxin Group | Polytrim Group
Number analyzed (Participants) | 28 | 31
participants | 22 | 19

ADVERSE EVENTS:
Arm/Group | Moxifloxacin Treatment Group | Polytrim Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 0/62 | 0/62

LIMITATIONS AND CAVEATS:
No adverse events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No